CLINICAL TRIAL: NCT03905486
Title: The Efficacy of Pregabalin as a Monotherapy Versus Combined Pregabalin and Milnacipran in the Management of Fibromyalgia.
Brief Title: Efficacy of Pregabalin Versus Combined Pregabalin and Milnacipran in Fibromyalgia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yousra Hisham Abdel Fattah (Other)
Responsible Party: Sponsor-Investigator, Yousra Hisham Abdel Fattah, Principle investigator, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0303417
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Fibromyalgia, Primary
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- G1: patients will receive pregabalin (Active Comparator): pregabalin as a mono-therapy will be administered in increment doses for 3 months
  Interventions: Drug: Pregabalin 300mg
- G2: patients will receive pregabalin and milnacipran (Active Comparator): pregabalin and milancipran as a combination therapy will be administered in increment doses for 3 months
  Interventions: Drug: Combined pregabalin 300mg and milancipran 100mg

INTERVENTIONS:
Drug: Pregabalin 300mg — Group 1: will receive pregabalin as a monotherapy. Pregabalin will be administered according to the treatment recommendations for fibromyalgia in the package insert [Pfizer Inc., 2012] starting by 50 mg twice daily increasing to 300 mg twice daily according to the efficacy and tolerability for 3 months.
  Arms: G1: patients will receive pregabalin
Drug: Combined pregabalin 300mg and milancipran 100mg — Group 2: will receive a combined pregabalin and milancipran. Pregabalin will be administered as group 1, while milancipran will be administered according to the treatment recommendations for fibromyalgia, starting by 50 mg once daily for 1 week then increased to reach 100 mg daily (50 mg twice daily) based on efficacy and tolerability for 3 month.
  Arms: G2: patients will receive pregabalin and milnacipran

SUMMARY:
Diagnosis of fibromyalgia is complex and treatment options are limited. Pharmacological management of fibromyalgia is mainly centered on the central nervous system. In particular there is robust evidence for the use of tricyclic antidepressants (e.g., amitriptyline), anti-convulsants such as gabapentin or pregabalin and agents from the serotonin norepinephrine reuptake inhibitor (SNRI) family such as milnacipran. Aim of the work: To compare the efficacy of pregabalin agent (averopreg) alone versus combined pregabalin and serotonin norepinephrine reuptake inhibitor (milnacipran) in the management of fibromyalgia.

DETAILED DESCRIPTION:
Subjects: The study will include 50 patients diagnosed as having fibromyalgia according to the ACR 2010 Fibromyalgia diagnostic criteria.

Methods: Patients will be classified into two groups:

1) Group 1: Patients will receive pregabalin as a monotherapy and the doses will be administered according to the treatment recommendations for fibromyalgia in the package insert, starting by 50mg twice daily increasing to 100 mg twice daily within 1 week based on efficacy and tolerability.

7) Group 2: Patients will receive combined pregabalin and milnacipran and the doses will be administered according to the treatment recommendations for fibromyalgia in the package insert, starting by 50mg twice daily increasing to 100 mg twice daily within 1 week for the pregabalin and starting by 12.5 mg increasing gradually to reach 100 mg daily of milnacipran based on efficacy and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* diagnosed as fibromyalgia according to the 2016 revision to the 2010/2011 fibromyalgia diagnostic criteria

Exclusion Criteria:

* Patients with major medical disorders or uncontrolled medical conditions
* Patients with recent myocardial infarction or stroke,
* Patients with active liver disease,
* Patients with renal impairment (creatinine clearance < 60 ml/min),
* Patients with documented autoimmune disease,
* Patients with severe chronic obstructive pulmonary disease,
* Patients with unstable diabetes,
* pregnancy or breastfeeding patients
* Patients with exposed to any investigational drug within the past 6 months

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females
Enrollment: 58 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
fibromyalgia impact questionnaire (FIQ) | 3 months
  assesses the overall functional ability and the impact of fibromyalgia on the patients life, with a range from 0-100, 0 indicating no functional impairment or effect of the disease on the patients life and 100 indicating a very bad and tremendous effect of fibromyalgia on the patients life
visual analogue scale (VAS) for pain | 3 months
  assesses the overall pain of fibromyalgia on a 100 mm pain scale with 0 indicating no pain and 100 indicating the worst pain ever

SECONDARY OUTCOMES:
Leeds sleep evaluation questionnaire | 3 months
  The four aspects of sleep around which the questionnaire is devised (Getting to sleep, GTS; Quality of sleep, QOS; Awakening from sleep, AFS; Behaviour following wakefulness, BFW), and assessing the effect of medication on the quality of sleep each question is a 100 mm line that the patient marks, 0 meaning very bad effect or worsening in sleep pattern, 50 meaning no improvement what so ever with no deterioration and 100 meaning excellent improvement in the sleep pattern

CONTACTS AND LOCATIONS:
Overall Officials: Yousra H Abdel-Fattah, Principal Investigator — Alexandria University Faculty of Medicine
Locations (1):
- Alexandria University, Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No